CLINICAL TRIAL: NCT05410678
Title: Safety And Efficacy Results of Percutaneous Renal Stent Implantation in Patients With Acute Coronary Syndrome With Ectatic and Aneurysmatic Coronary Arteries
Brief Title: Safety And Efficacy Results of Percutaneous Renal Stent Implantation in Ectatic and Aneurysmatic Coronary Arteries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Prof. Dr., Bursa Postgraduate Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBU Bursa PH
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- renal stent group (Experimental): Acute coronary patients treatment with renal stent
  Interventions: Drug: Renal stent
- BMCS group (Active Comparator): Acute coronary patients treatment with bare-metal stent
  Interventions: Drug: Renal stent

INTERVENTIONS:
Drug: Renal stent — renal stent implantation in ectatic/aneurysmatic coronary arteries
  Other Names: Renal stent for coronary artery

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of renal stents implanted in ectatic/aneurysmatic coronary arteries.

DETAILED DESCRIPTION:
In total, 18 patients (renal stent group) who underwent renal stent implantation in ectatic/aneurysmatic coronary arteries requiring percutaneous coronary intervention (PCI) and 45 patients who underwent large-sized bare metal coronary stent (BMCS) implantation (BMCS group) at our centre between 2015 and 2020 were included in the study. Control coronary angiography (CAG) was performed during the follow-up of these patients, and angiography-guided quantitative measurements were performed during PCI. The primary endpoints were myocardial infarction and cardiovascular mortality, and the secondary endpoints were restenosis and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome patients

  * 18 year age
* ectatic/aneurysmatic coronary arteries

Exclusion Criteria:

* Patients who underwent elective procedures,
* experienced unsuccessful attempts
* referred to surgical revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
primary endpoints | 2 year
  Rate of myocardial infarction and cardiovascular mortality

SECONDARY OUTCOMES:
secondary endpoints | 2 year
  Rate of restenosis and all-cause mortality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camci S, Ari H, Sunbul A, Ari S, Melek M, Bozat T. Safety and efficacy results of percutaneous renal stent implantation in patients with acute coronary syndrome with ectatic and aneurysmatic coronary arteries. Postgrad Med. 2024 Jan;136(1):95-102. doi: 10.1080/00325481.2024.2313447. Epub 2024 Feb 5. PMID 38299468